CLINICAL TRIAL: NCT00697931
Title: Study to Compare the Immunogenicity and Reactogenicity of GSK Biologicals; (Previously SmithKline Beecham Biologicals') MPL-Adjuvanted Recombinant Hepatitis B Vaccine With That of Engerix™-B in an Adult Non-Responder Population
Brief Title: Immunogenicity and Reactogenicity of MPL Adjuvanted Recombinant Hepatitis B- Vaccine and Engerix™-B in Adult Non-Responders
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Isabelle Harpigny, GSK
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 208129/021
Record Dates: First submitted 2008-06-12; First posted 2008-06-16 (Estimated); Last update posted 2008-06-16 (Estimated); Status verified 2008-06

CONDITIONS: Hepatitis B
Keywords: Hepatitis B; Engerix™-B; Recombinant Hepatitis B vaccine; Adjuvant
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Group A (Experimental)
  Interventions: Biological: Recombinant MPL- adjuvanted hepatitis B vaccine
- Group B (Active Comparator)
  Interventions: Biological: Engerix™-B

INTERVENTIONS:
Biological: Recombinant MPL- adjuvanted hepatitis B vaccine — Intramuscular injection, 3 doses
  Arms: Group A
Biological: Engerix™-B — Intramuscular injection, 3 doses
  Arms: Group B

SUMMARY:
The purpose of this study is to compare the immunogenicity and reactogenicity of the adjuvanted recombinant hepatitis B vaccine with that of Engerix™-B when both are injected according to a three dose schedule (0, 1, 6 months) in an adult non-responder population

DETAILED DESCRIPTION:
At the time of conduct of this study, the sponsor GlaxoSmithKline was known by its former name SmithKline Beecham

ELIGIBILITY:
Inclusion Criteria:

* Age: older than 18 years of age.
* Documented non-responders 2 to 5 months after having received 4 doses of a hepatitis B vaccine
* Good physical condition as established by clinical examination and history taking at the time of entry.
* Female participants who are at risk to become pregnant will be on a contraceptive programme if necessary during the study period.
* Written informed consent obtained from the subjects

Exclusion Criteria:

* Positive at screening for anti-HBV antibodies
* Elevated serum liver enzymes.
* History of significant and persisting hematologic, hepatic, renal, cardiac or respiratory disease.
* Any acute disease at the moment of entry.
* Chronic alcohol consumption.
* Hepatomegaly, right upper quadrant abdominal pain or tenderness.
* Any chronic drug treatment, including any treatment with immunosuppressive drugs, which in the investigator's opinion, precludes inclusion into the study.
* History of allergic disease likely to be stimulated by any component of the vaccine.
* Simultaneous participation in any other clinical trial.
* Previous vaccination with an MPL containing vaccine.
* Administration of immunoglobulins 6 months before and during the whole study period
* Vaccination one month before and one month after each dose of the study vaccine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 1997-05; Primary Completion 1998-06 (Actual); Study Completion 1998-06 (Actual)

PRIMARY OUTCOMES:
Anti-HBs antibody concentrations | At month 7

SECONDARY OUTCOMES:
Anti-HBs antibody concentrations | At months 2, 6, 7 and 12
Occurrence and intensity of solicited local symptoms | 4-day follow-up after vaccination
Occurrence, intensity and relationship of solicited general symptoms | 4-day follow-up after vaccination
Occurrence, intensity and relationship to vaccination of unsolicited symptoms | Within 30 days after vaccination
Incidence of serious AEs | Throughout the entire study up to and including 30 days after the last vaccination
Cell mediated immunity | At months 0, 2, 6, 7, 12

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Clinical Trials Call Center, Leuven, Belgium